CLINICAL TRIAL: NCT01766752
Title: An Open, Single-centre, Non-controlled Feasibility Study of the Performance of a Tablet Based Workflow and Decision Support System With Incorporated Software Algorithm Used for Glycaemic Management in Non-critically Ill Patients With Type 2 Diabetes at the General Ward
Brief Title: Performance of a Tablet Based Workflow and Decision Support System With Incorporated Software Algorithm Used for Glycaemic Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Medical University of Graz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClinDiab-03
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- GlucoTab System (Experimental): Investigational system: GlucoTab system supports the glycaemic management of non-critically ill patients with type two diabetes at the general ward.
  Interventions: Device: GlucoTab System
- no intervention (No Intervention): standard care

INTERVENTIONS:
Device: GlucoTab System — Tablet based workflow and decision support system with incorporated software algorithm (GlucoTab) used for glycaemic management in non-critically ill patients with type 2 diabetes at the general ward
  Arms: GlucoTab System

SUMMARY:
Objective: To investigate the performance (safety) of the GlucoTab system for glycaemic management in non-critically ill patients with type 2 diabetes at the general ward

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged 18 - 90 years (both inclusive)
* Type 2 diabetes treated with diet, oral agents, non-insulin injected anti-diabetic medicine, insulin therapy or any combination of the four

Exclusion Criteria:

* Impaired renal function (serum creatinine ≥3.0mg/dL)
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient
* Pregnancy
* Any mental condition rendering the patient incapable of giving his consent
* Terminally ill patients
* Participation in a trial within 3 months prior to this trial
* Known or suspected allergy to insulin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percentage of actions the system supports either to capture BG values or provide insulin dose suggestions according to the REACTION algorithm. | duration of hospital stay (maximum three weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Schaupp L, Donsa K, Neubauer KM, Mader JK, Aberer F, Holl B, Spat S, Augustin T, Beck P, Pieber TR, Plank J. Taking a Closer Look--Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients with Type 2 Diabetes Mellitus Under Basal-Bolus Insulin Therapy. Diabetes Technol Ther. 2015 Sep;17(9):611-8. doi: 10.1089/dia.2014.0343. Epub 2015 Apr 30. PMID 25927357